CLINICAL TRIAL: NCT01331980
Title: Bone Microarchitecture at the Radius: a Pilot Comparison Between Children With Cystic Fibrosis and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 113442
Record Dates: First submitted 2011-03-15; First posted 2011-04-08 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; bone
MeSH Terms: conditions — Cystic Fibrosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples will be frozen and assayed together.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cystic fibrosis: children aged 6-12 years of age and Tanner stage 1 with a diagnosis of cystic fibrosis
  Interventions: Device: Peripheral quantitative computed tomography (pQCT); Device: Dual X-ray absorptiometry (DXA)
- healthy controls: children ages 6-12 years and Tanner stage 1 without cystic fibrosis or other chronic disease that affects bone health
  Interventions: Device: Peripheral quantitative computed tomography (pQCT); Device: Dual X-ray absorptiometry (DXA)

INTERVENTIONS:
Device: Peripheral quantitative computed tomography (pQCT) — A pQCT scan of the non-dominant radius at the 4% and 65% sites will be conducted at a single study visit
  Other Names: Stratec XCT 2000 series pQCT
Device: Dual X-ray absorptiometry (DXA) — A total body DXA scan will be conducted at a single study visit
  Other Names: Hologic QDR 4500A

SUMMARY:
Cystic fibrosis (CF) affects an estimated 30,000 people in the United States and is caused by a mutation in the gene encoding a protein called CF transmembrane regulator (CFTR). The hallmarks of CF are recurrent pulmonary exacerbations and declining pulmonary function. However, there are other problems in CF that affect both health and quality of life. These include CF related diabetes, liver disease, and bone disease. The median age of survival for patients with CF has been increasing steadily and is currently more than 37 years. With this improvement in life expectancy, it has become increasingly important to address the long-term complications of CF.

Currently, patients with CF are evaluated annually for bone disease with dual X-ray absorptiometry (DXA), and screening usually starts at age 12. However, this may not be sufficient to detect early bone changes that may impact fracture risk. Furthermore, bone disease in children may manifest earlier than adolescence, which would suggest that screening should start at an earlier age in these vulnerable patients. The following study is therefore proposed to examine the potential role of peripheral quantitative computed tomography (pQCT) as a screening approach for bone disease in children with CF. The investigators expect to find bone problems by pQCT but not DXA.

DETAILED DESCRIPTION:
This is a single-center study

1. STUDY OBJECTIVES

   1.1 Primary Objective Compare bone measurements (by pQCT of the radius and DXA scan of the lumbar spine and total body) in children with CF 6-12 years of age to healthy children. Measurements by pQCT to be compared will include cortex width, trabecular bone mineral density (BMD), and volumetric BMD. Measurements by DXA to be compared will include total body bone mineral density and lumbar spine (L1-L4) BMD.

   1.2 Secondary Objectives Compare Z-scores of pQCT parameters to Z-scores of BMD as measured by DXA in children with CF 6-12 years of age. The Z-scores for each CF subject for pQCT measurements (cortex width, trabecular BMD, volumetric BMD) and DXA measurements (total body BMD and lumbar spine BMD) will be compared.

   Compare correlation of pQCT parameters and BMD as measured by DXA to markers of bone turnover and inflammation (serum propeptide of type I collagen (PICP), total serum deoxypyridinoline, C-reactive protein (CRP), interleukin 6 (IL-6), and tumor necrosis factor (TNF)-alpha) in children with CF 6-12 years of age and healthy controls. As an exploratory specific aim, the correlation between these serum markers and the bone measurements in Specific Aim 1 will be evaluated.
2. BACKGROUND AND RATIONALE

Cystic fibrosis (CF) affects an estimated 30,000 people in the United States1 and is caused by a mutation in the gene encoding a protein called CF transmembrane regulator (CFTR). This protein functions as a chloride channel in epithelial cells of multiple organ systems. The mutation results in a dysfunctional or absent CFTR channel and a decrease in chloride secretion, which ultimately results in increased viscosity of secretions. Children with CF are less able to clear pulmonary secretions and become colonized with bacterial pathogens that regularly cause exacerbation of lung disease. The hallmarks of CF are recurrent pulmonary exacerbations and declining pulmonary function. Respiratory failure is the cause of death in more than 90% of people with CF. However, there are also extrapulmonary manifestations of CF that affect both health and quality of life. These include CF related diabetes, liver disease, and bone disease. The median age of survival for patients with CF has been increasing steadily and is currently more than 37 years.1 With this improvement in life expectancy, it has become increasingly important to address the long-term complications of CF.

There is a high prevalence of osteopenia and osteoporosis among both adult and pediatric patients with CF and this steadily increases with age. There is also an associated increase in fracture rate and kyphosis in adults. Studies evaluating fracture risk in children with CF have generated mixed results. Henderson et al reported an increased rate of fracture in girls with CF, but not boys, in comparison to healthy controls. A more recent study by Rovner et al showed no increase in fracture risk among children with mild to moderate lung disease. Bisphosphonates have been used to treat osteopenia and osteoporosis in adults with CF and clinical trials have shown that there is an increase in bone mineral density (BMD) with therapy. However, there is no published data demonstrating a reduced fracture rate with bisphosphonate therapy. Furthermore, there is currently no consensus on how to treat osteopenia or osteoporosis in children with CF other than to ensure adequate nutrition and vitamin D levels. Although CF bone disease is considerably more prevalent in the adults than in children, screening for bone disease must be addressed in childhood to maximize peak bone mass and potentially minimize bone related disease in these patients.

Biochemical markers of bone turnover may be used to evaluate derangements in bone formation and/or resorption. Studies conducted in CF patients have shown in general a decrease in markers of bone formation and increase in markers of bone resorption. Conway et al reported correlation between markers of bone turnover and both spinal and total body BMD; however, no studies have evaluated whether bone turnover markers correlate with pQCT parameters. Serum PICP is a peptide cleaved from the carboxy-terminal end of collagen type I and is a marker of bone formation. Deoxypyridinoline is a cross-linking amino acid that is released from the bone matrix by resorption, and thus is a marker of bone resorption.

The etiology of bone disease in patients with CF is multifactorial and contributing factors include poor nutrition, decreased activity levels, poor absorption of vitamin D, chronic inflammation, and therapy with corticosteroids. Multiple studies have correlated BMD with clinical factors such as lung function, nutritional status, inflammation markers, clinical score, and frequency of antibiotic courses. Studies evaluating the relationship between inflammation markers and bone in CF patients have been somewhat mixed, although in general have shown an inverse relationship between inflammation and BMD, and a direct correlation between inflammation and increased bone resorption markers. Inflammation markers evaluated have included both acute-phase cytokines such as IL-6 and TNF-alpha, and the general marker CRP. There is some evidence that CFTR is expressed in bone cells such as osteoclasts, osteoblasts, and osteocytes, suggesting the potential for a bone phenotype in patients with CF. Most studies utilize DXA and demonstrate reduced BMD in patients with CF that is usually detectable starting in adolescence. Low BMD is nearly universal among adults with CF; however, results from studies evaluating BMD in children with CF have been variable.

A study conducted in adolescents and young adults with CF utilized pQCT to evaluate bone geometry of the radius. Although BMD was normal for these subjects, pQCT data indicated that the subjects had a reduced cortical thickness. Reduced cortical thickness has been shown in cadaveric studies to be predictive of mechanical strength. Currently, patients with CF are evaluated annually for bone disease with DXA, and screening usually starts at approximately age. However, the above study suggests that this approach may not be sufficient to detect early bone changes that may impact fracture risk. Furthermore, bone disease in children may manifest earlier than adolescence, which would suggest that screening should start at an earlier age in these vulnerable patients. The following study is therefore proposed as a translational pilot study to examine the potential role of pQCT as a screening approach for bone disease in children with CF. The investigators expect to find bone deficits by pQCT but not DXA, and better correlation of inflammation and bone turnover markers with pQCT measurements than with DXA measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF by sweat test and/or genotyping for CF subjects (for CF group only)
* 6-12 years of age at time of study visit
* Body mass index of at least the 3rd percentile
* Tanner stage 1

Exclusion Criteria:

* Body mass index (BMI) greater than the 95th percentile
* Recent fracture (within the past 6 months)
* Lung transplant recipient
* Current pulmonary exacerbation or current infection
* History of bisphosphonate or growth hormone therapy (in the past 5 years)
* Glucocorticoid therapy within the past 6 months
* Severe pulmonary dysfunction (forced expiratory volume in 1 second < 40% predicted) if subjects are performing spirometry
* Concomitant disease known to cause bone disease (e.g. chronic kidney disease, CF-related diabetes)
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants for the cystic fibrosis (CF) group will be recruited from the pulmonary clinic at Arkansas Children's Hospital. Healthy controls will be recruited from Arkansas Children's Hospital outpatient clinics and the community.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Peripheral quantitative computed tomography (pQCT) - cortex width | Day 1
  pQCT scan of the non-dominant radius at the 4% and 65% sites will be conducted and parameters will include cortex width, trabecular bone mineral density (BMD), and total BMD
pQCT parameters - trabecular BMD | Day 1
  pQCT scan of the non-dominant radius at the 4% and 65% sites will be conducted and parameters will include cortex width, trabecular BMD, and total BMD
pQCT parameters - total BMD | Day 1
  pQCT scan of the non-dominant radius at the 4% and 65% sites will be conducted and parameters will include cortex width, trabecular BMD, and total BMD.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine O'Brien, PharmD, Principal Investigator — University of Arkansas for Medical Sciences and Arkansas Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States